CLINICAL TRIAL: NCT05880342
Title: Investigating Fundamental Mechanisms of Mental and Physical Fatigue Using Neurotransmitter Reuptake Inhibitors and Electroencephalography: a Randomized Counterbalanced Crossover Trial
Brief Title: The Role of the Brain in Mental and Physical Fatigue
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Science and Research Centre Koper (Other)
Responsible Party: Principal Investigator, Yahaira Laurisa Arenales Arauz, Yahaira Laurisa Arenales Arauz, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: G095422N
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Reboxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mental fatigue group (Other)
  Interventions: Drug: Reboxetine Pill; Drug: Methylphenidate Oral Product
- Physical fatigue group (Other)
  Interventions: Drug: Reboxetine Pill; Drug: Methylphenidate Oral Product
- Combined group (Other)
  Interventions: Drug: Reboxetine Pill; Drug: Methylphenidate Oral Product

INTERVENTIONS:
Drug: Reboxetine Pill — 8 mg
Drug: Methylphenidate Oral Product — 20 mg

SUMMARY:
The goal of this clinical trial is to determine the role of brain neurotransmission in the onset of fatigue, identify the brain areas involved, and determine how brain activity and neuromuscular efficiency changes during onset of fatigue. Three different experimental studies (physical fatigue, mental fatigue and combined) will be performed with a randomized, single-blinded, placebo controlled, counter-balanced, cross-over design.

The objectives of the projects are as follows:

* To experimentally assess the role of a dopamine, and a noradrenalin reuptake inhibitor in the onset of exercise-induced fatigue
* To identify changes in brain activation associated with altered PF and fatigue perception
* To experimentally assess the effect of a NA or DA reuptake inhibitor on MF, brain activation and the sources of changes in brain activation
* To experimentally assess the role of brain neurotransmitters (DA, NA) in the interaction between mental and PF from a neurophysiological perspective.

Participants will be healthy young adults. In each study, they will start with a familiarization trial followed by two experimental trials and one control trial with a randomized treatment order. At each visit, different drugs will be administered to elicit different neurotransmitter response. The trials will be performed at the MFYS exercise lab (BLITS, VUB campus Etterbeek, Boulevard General Jaques 271, 1050 Elsene (Brussels)).

Depending on the type of study they are participating in, participants will perform three distinct tasks:

* In the first experimental study participants will perform a 60-min Stroop Task to elicit mental fatigue.
* In the second experimental study participants will perform a knee-extension exercise until exhaustion to elicit physical fatigue.
* In third experimental study participants will first preform a mental fatiguing task (Stroop taks) followed by physical fatigue task (knee extension).

While participants will perform above mentioned task their EEG signal and heart rate will be measured. At the same time, participants will report on their subjective feeling of fatigue during these tasks. In addition, all participants will be administered cognitive tasks before and after the study, along with questionnaires. In the second and third experiments, tensiomyography and electromyography will also be recorded from the quadriceps muscle of the leg used for knee extension.

Researchers will compare physiological and behavioural changes in response to specific neurotransmitter drug to answer the main question: what the role of a DA and a NA reuptake inhibitor on the onset of mental and physical fatigue is.

ELIGIBILITY:
Inclusion Criteria:

* Healthy trained individuals (exercises at least 1x per week, no neurological, cardiovascular internal or musculoskeletal disorders of any kind)
* No use of chronic or occasional prescribed medication (except for contraceptives)
* Non-smoker

Exclusion Criteria:

* Injuries of any kind in the past 6 months
* Pregnancy
* Specific food or drink allergies (e.g. lactose and/or gluten intolerance)
* Suffering from a chronic health condition (could be neurological, cardiovascular, internal and musculoskeletal)
* Participating in any concomitant care or research trials
* History of suffering from any mental/psychiatric disorders:

Suffering from a higher risk of burn out, indicated by a total score of more than 2.59 on the Burn out assessment tool (BAT) Suffering from high general fatigue, indicated by a score of more than 57 on the Multidimensional fatigue inventory (MFI) Suffering from depression, indicated by a score of more than16 on the Beck depression inventory-II (BDI-II)

* Use of medication Chronic use with an exception for contraceptives Prescribed medication in between or before trials Use of non-prescribed occasional medication 24 hours prior each trial
* Use of caffeine and heavy efforts 24 hours prior each trial
* Suffering from colour vision deficiencies
* Not eating a standardized meal, the morning of each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of repetitions | 30 minutes
  Number of repetitions during knee extension task
Electroencephalography (spectral analysis) | 80 minutes
  measurement of cortical activity with 64 channels (spectral density in alpha, beta, gamma, delta, theta)
Electroencephalography (event related potentials) | 80 minutes
  measurement of cortical activity with 64 channels (event related potentials)
Electromyography | 60 minutes
  Target muscles are rectus femoris and vastus lateralis (median frequency)
Accuracy | 60 minutes
  Accuracy of correct answers during Stroop task
Reaction time | 60 minutes
  Reaction time for answers during Stroop task

SECONDARY OUTCOMES:
Perceived stress scale questionnaire (PSS-10) | 5 minites
  Result is the score of the questionnaire (may 40 points)
the international physical activity questionnaire short form (IPAQ-SF) | 2 minutes
  Result is the score of the questionnaire
The Brunel Mood Scale (BRUMS) | 5 minutes
  Result is the score of the questionnaire (each subscale max 0-16)
Motivation with visual analog score (Moti-VAS) | 1 minute
  Result is the score between 0 and 100
The National Aeronautics and Space Administration Task Load Index (NASA-TLX) | 3 minutes
  Result is the score of the questionnaire
Subjective feeling of Mental Fatigue with visual analog score (M-VAS) | 1 minute
  Result is the score between 0 and 100
Subjective feeling of physical fatigue with visual analog score (P-VAS) | 1 minute
  Result is the score between 0 and 100
Karolinska Sleepiness Scale (KSS) | 5 minutes
  Result is the score of the questionnaire (max 24)
Internal load of the physical performance (CR100 RPE) | 30 minutes
  Result is the score between 0 and 100
Heart Rate | 60 minutes
  continuously assessed by using the POLAR H10 sensor
Lactate concentration | 5 minutes
  blood lactate will be measured at the beginning and end of the trial at the finger tip of the participant (unit = mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels Labo voor Inspanning & Topsport U-residence, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arauz YLA, Mali A, Lathouwers E, Habay J, Fortes LS, Meeusen R, Marusic U, De Pauw K, Roelands B. Distinct Roles of Dopamine and Noradrenaline in Physical Fatigue. Eur J Sport Sci. 2026 Feb;26(2):e70119. doi: 10.1002/ejsc.70119. PMID 41601207